CLINICAL TRIAL: NCT04869683
Title: Biocollection in Patients With Myelodysplastic Syndrome (P-MDS)
Brief Title: Biocollection in MyeloDysplastic Syndrome (P-MDS)
Acronym: P-MDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 29BRC20.0228
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Myelodysplastic Syndromes; Myelodysplastic Anemia; Myelodysplastic Syndrome With Isolated Del(5Q); Myelodysplastic Syndrome With Ring Sideroblasts; Acute Myeloid Leukemia With Multilineage Dysplasia; Chromosome Abnormality
Keywords: MDS; 5q deletion; ring sideroblasts; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Chromosome 5q Deletion Syndrome; Chromosome Aberrations

STUDY DESIGN:
Intervention Model Description: Health services research and follow up DMS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDS follow up (Other): it is a description MDS patients study
  Interventions: Other: description of MDS pzatient cohort

INTERVENTIONS:
Other: description of MDS pzatient cohort — description of MDS patient cohort

SUMMARY:
Myelodysplastic syndromes (MDS) are chronic myeloid hemopathies characterized by ineffective hematopoiesis (with peripheral cytopenias) and which contrast with a marrow of normal richness. MDS is considered one of the four most common blood diseases. The incidence is estimated at 4,059 cases / year in 2012 with an average age of 78 years in men and 81 years in women (INCA report, Cancers in France in 2015). The incidence increases with lengthening of the lifespan. The main risk of MDS is transformation to acute leukemia in 30 to 40% of cases. Treatment options depend on clinical, hematologic and chromosomal abnormalities. The prognosis is considered to be at low or high risk of developing acute leukemia. This distinction will therefore have an impact on the therapeutic solution (s). MDS exhibit clinical, morphological and genetic heterogeneity. It is therefore necessary to form subgroups of patients to better understand the physiopathogenesis of this pathology. The constitution of a biocollection will make it possible to search for clinical and biological prognostic markers in order to identify patients progressing to acute myeloid leukemia.

DETAILED DESCRIPTION:
The objective of the biocollection is to respond to 3 scientific projects in MDS :

Project 1: splicing anomalies in MDS with SF3B1 mutations : About 95% of the coding genes in humans are subjected to alternative splicing, a complex, highly regulated mechanism that diversifies the proteome by defining multiple proteins from a single gene. Deregulation of splicing is observed in many cancers and hemopathies (review Yoshida et al., 2014), especially in myelodysplastic syndromes More than half of MDS patients present an acquired mutation in a gene involved in the splicing of pre -RNA messengers. The SF3B1 gene (splice factor 3B subunit 1), which encodes a protein involved in the recognition of 3 'splice sites is the most frequently mutated gene in SMDs, at a frequency of 20-28% MDS, and up to 85% of myelodysplastic syndromes with crowned sideroblasts (Yoshida et al., 2011, Papaemmanuil et al., 2011). The functional consequences of the splicing abnormalities thus generated on the pathophysiology of MDS are far from clear. The transcriptome analyzes (by RNA-seq) carried out recently in various acquired pathologies that the most frequent variants of the SF3B1 gene lead to the formation of aberrant transcripts by the use of a 3 ' cryptic splicing site. The investigators seek to study the functional implications of SF3B1 mutations found in MDS patients in particular on the formation of sideroblasts in the crown. The investigators want to identify, by RNAseq, the aberrant junctions specifically expressed in the cells of MDS patients with mutated SF3B1, and which would affect transcripts of genes involved in iron metabolism or its regulation. For this, the investigators will use the cells obtained from the marrow of SMD SF3B1WT patients versus SF3B1K700E and collected in the Chromosomal Genetics laboratory, site of the CRB of the CHRU of Brest. The investigators will then analyze the functional repercussions associated with the presence of these aberrant junctions on the cells in culture of these same patients (detection of certain proteins, enzymatic analyzes, etc.). The collection of biological and clinical data from these patients of interest is essential for the interpretation of the results. This project is part of a more global approach to the study of the various splicing anomalies in this pathology.

Project 2: splicing abnormalities in MDS with chromosomal abnormalities as 5q deletion : Chromosome 5 deletions are the most frequent structural abnormalities in MDS and constitute a good prognostic entity if isolated or associated with an anomaly and poor prognosis if associated with more than 3 chromosomal abnormalities. Two genes located on chromosomes 5 encode proteins of a complex involved in the splicing of pre-messenger RNAs: the RBM22 gene (RNA Binding Motif Protein 22) and the SLU7 gene (SLU7 Homolog Splicing Factor).

The investigators want to identify subgroups of patients with loss of these 2 genes or loss of RBM22 and conservation of SLU7. Does the loss of one or both genes play a role in the pathophysiogenesis of MDS with chromosome deletions and is it associated with worsening of the disease? Understanding these mechanisms could also have an impact on the therapeutic management of this pathology.

The study of these chromosomal abnormalities associated with splicing abnormalities in MDS for the chromosomal genetics laboratory both from a diagnostic and research perspective. Several works carried out have given rise to numerous scientific publications with an international reading committee for several years.

Project 3: Evolution of MDS in acute myeloid leukemia (AML) More than one third of patients with MDS progress to AML. The investigators want to focus on this group of patients and understand the clonal architecture of their malignant cells to detect new predictive markers of indolent or rapid disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Major
* patient with or suspected of myelodysplastic syndrome (WHO definition) at diagnosis and/or during follow-up, which is managed at the level of the Cancer-Hematology Institute of the Brest CHRU
* Presence of biological material collected within the CRB
* Patient's consent obtained

Exclusion Criteria :

* Minor and pregnant woman
* Lack of biological material collected within the CRB
* Refusal to participate: lack of consent - Unable to consent
* Patient under judicial protection: guardianship, curatorship ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2032-10-19 (Estimated); Study Completion 2032-10-19 (Estimated)

PRIMARY OUTCOMES:
Cohort MDS: epidemiologic MSD study | five years
  MDS study in collecting data

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Douet-Guilbert, MD,PhD, Principal Investigator — CHRU Brest
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement